CLINICAL TRIAL: NCT04026139
Title: Elastic Band Resistance Exercise on Glycated Haemoglobin and Muscle Strength, Balance, and Physical Function in Patients With Comorbid Type 2 Diabetes Mellitus and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Mei Chen (Other)
Responsible Party: Sponsor-Investigator, Shu-Mei Chen, ChangGungMH, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201700009B0D001
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Elastic Band Resistance Exercise With Comorbid Type 2 Diabetes Mellitus and Knee Osteoarthritis
Keywords: home-based exercise, resistance band, cartilage degeneration, glycated haemoglobin control, diabetes mellitus
MeSH Terms: conditions — Osteoarthritis, Knee; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Design: Randomised controlled trial. Participants: Seventy patients diagnosed with T2DM together with knee OA. Intervention: Patients in the experimental and control group were instructed by clinical staff to perform home-based exercises and followed up through phone calls. The experimental group performed exercises using an elastic resistance band with 10 repetitions/set × 5 sets/day × 3 days/week. The control group underwent active joint range-of-motion exercises and isometric contraction exercises. The intervention regimens lasted 12 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients in the experimental and control group were instructed by clinical staff to perform home-based exercises and followed up through phone calls. The experimental group performed exercises using an elastic resistance band with 10 repetitions/set × 5 sets/day × 3 days/week.
  Interventions: Other: Elastic Band Resistance Exercise
- control group (Active Comparator): The control group underwent active joint range-of-motion exercises and isometric contraction exercises.
  Interventions: Other: active joint range-of-motion exercises and isometric contraction exercises

INTERVENTIONS:
Other: Elastic Band Resistance Exercise — Patients in the experimental and control group were instructed by clinical staff to perform home-based exercises and followed up through phone calls. The experimental group performed exercises using an elastic resistance band with 10 repetitions/set × 5 sets/day × 3 days/week.
  Arms: experimental group
Other: active joint range-of-motion exercises and isometric contraction exercises — The control group underwent active joint range-of-motion exercises and isometric contraction exercises. The intervention regimens lasted 12 weeks.
  Arms: control group

SUMMARY:
Whether elastic band resistance exercise (EBRE) as a home-based rehabilitation routine can control the glycated heamoglobin (HbA1c) level and improve the muscle strength, dynamic balance, and physical function in older patients with comorbid T2DM and knee OA?

DETAILED DESCRIPTION:
Design: Randomised controlled trial. Participants: Seventy patients diagnosed with T2DM together with knee OA. Intervention: Patients in the experimental and control group were instructed by clinical staff to perform home-based exercises and followed up through phone calls. The experimental group performed exercises using an elastic resistance band with 10 repetitions/set × 5 sets/day × 3 days/week. The control group underwent active joint range-of-motion exercises and isometric contraction exercises. The intervention regimens lasted 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study were as follows: age between 60 and 70 years; comorbid T2DM and knee OA diagnosed by a physician; and Kellgren and Lawrence (K&L) grade <3 based on the findings of plain radiographs.

Exclusion Criteria:

* Exclusion criteria were as follows: inability to perform any self-activity; DM with complications, such as lower extremity neuropathy, retinopathy, stroke, foot wounds, or amputations; K&L grade >3, hip or knee arthroplasty; history of myocardial infarction; uncontrolled liver and kidney disease; and uncontrolled hypertension.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
HbA1c level | up to 12 weeks of intervention
  follow blood glucose cotrol
WOMAC physical function subscale scores | up to 12 weeks of intervention
  follow osteoarthritis physical function
30-s chair stand test [CST] | up to 12 weeks of intervention
  follow low leg muscle strength
3-m timed up and go test [TUG] | up to 12 weeks of intervention
  follow dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Jen Chang, Study Director — Kaohsiung Medical University Department of Sports Medicine professor
Locations (1):
- Shu-Mei Chen, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage, and then share with other researchers after publication.